CLINICAL TRIAL: NCT03246464
Title: Orthokeratology Contact Lenses for the Treatment of Myopia in a Group of Danish Children
Brief Title: Clinical Study Of Nearsightedness; TReatment With Orthokeratology Lenses (CONTROL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Ens Eyes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CONTROL
Record Dates: First submitted 2017-07-11; First posted 2017-08-11 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Myopia
Keywords: Contact lenses; Children; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Randomized controled clinical interventional trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-vision spectacles (Placebo Comparator)
  Interventions: Device: Single-vision spectacles
- Orthokeratology lenses (Active Comparator)
  Interventions: Device: Orthokeratology lenses

INTERVENTIONS:
Device: Orthokeratology lenses — Rigid gas permeable contact lenses
  Arms: Orthokeratology lenses
Device: Single-vision spectacles — Regular single vision spectacles
  Arms: Single-vision spectacles

SUMMARY:
Myopia is a common disease of the eye with increasing prevalence in the Western World as well as in South East Asia where 60-90% of the children are affected. High myopia is associated with an increasing risk of sight threatening complications such as retinal detachment, glaucoma, macular choroidal degeneration and myopic choroidal neovascularization. In myopia the eye is elongated compared to an emmetropic eye. If the elongation of the eye can be controlled the progression of myopia can be controlled. Asian studies have shown reduction in axial length growth by 36-46% in children using orthokeratology contact lenses (OKL). OKL are custom fit, form stable lenses. During sleep the cornea is reshaped creating an emmetropic vision during the day, so no glasses or contact lenses are needed. Twin and family studies have shown a high heritability for the development of myopia, and more than 40 genetic loci have been identified indicating that the effect of OKL in Asian children might not be the same in North European children which is why we want to execute a similar study on North European children.

Purpose:

1. Investigate if nightly wear of OKL reduces the progression of childhood myopia (change in axial length) in Danish children when compared to a control group using monofocal glasses.
2. Investigate the safety (Efron score) of OKL.
3. Investigate children's quality of life impact of refractive correction (questionnaire) using OKL compared to glasses.
4. Identify possible predictors for progression of myopia (AC/A ratio, peripheral defocus and higher order aberrations).

Method:

A randomized controlled 18 months prospective 1:1 study of a group of Danish children. 60 children will be included; 30 in each group. The participants will undergo several measurements reflecting the anatomy and function of the eye at baseline, 6, 12 and 18 month to evaluate the effect.

DETAILED DESCRIPTION:
Myopia is a common disease of the eye with increasing prevalence in the Western World as well as in South East Asia where 60-90% of the children are affected. A Danish study found that early debut of myopia is associated with a higher degree of myopia later on in life. Myopia may be corrected with spectacles, contact lenses or surgically, but despite this socio-economic burden, high myopia is associated with an increasing risk of sight threatening complications such as retinal detachment, glaucoma, macular choroidal degeneration and myopic choroidal neovascularization.

Myopia is a complex disease with a multi-factorial etiology. Twin studies and family studies have shown a high heritability for development of myopia, and more than 40 genetic loci have been identified. Outdoor activity seems to reduce the myopia progression. The shape of the eye may be of importance; axial growth makes the eye ellipsoidal which increase the peripheral defocus on the retina. Peripheral defocus has been suggested to induce further axial growth of the eyeball.

Accommodation is a significant covariant of near work and reading. A cross section study has shown a reduced precision in accommodation (A) on a near object combined with increased convergence (C) in myopic eyes. This increased AC/A ratio (dynamic) may be a predictor for myopia progression.

Interventions for reducing myopia progression have been many. The effects of progressive additional lenses, multifocal lenses and bifocal lenses have been limited. Anticholinergic eyedrops (Atropin 0.01%) significantly reduce the progression of myopia in Asian children by approximately 50% over a period of two years with limited side effects. Almost similar results have been found in Asian children using orthokeratology contact lenses (OKL) for reducing myopia progression.

OKL are custom fit, form stable lenses used during sleep. The lenses induce a temporal flattening of the cornea, which modify or eliminate refractive errors, leaving no need for glasses or contact lenses during daytime. OKL were introduced in the 1960 ́s, but with limited success due the lens material (PMMA) which was not gas-permeable. Decentration was also a problem making the effect variable and unpredictable. With new gas- permeable lens materials and computer assisted topographic measurements of the cornea, fitting of the lenses has been improved significantly, so that nightly wear is now standard treatment.

A clear-cut reduction in axial length growth in Asian children using OKL compared to single-vision spectacles (SVS) has been proofed in several studies. In these studies, which are very heterogeneous regarding design, reductions of 36-46% in axial length growth were found compared to a matched control group. Two European prospective cohort studies have investigated the effect of OKL compared to SVS in Spanish children. A reduction in axial growth of 32 % and 38% respectively was found. Side effects of OKL have been evaluated; in a meta-analysis from 2015, including 8 Asian and one of the European studies. Odds Ratio for side effects were 8.87 for the OK group compared to the control group, however all side effects were mild and disappeared after termination of the treatment.

Thus, a reduction in childhood myopia using OKL has been proofed in Asian children; however, weather similar result can be achieved in a group of children from Northern Europe is unknown. The influence of OKL on quality of life impact of refractive correction has never been investigated in a randomized trail. How OKL reduce the axial growth of the eye is unknown. The lenses induce multifocality and higher order aberrations in the cornea, which might change the peripheral defocus. A change in defocus has been suggested as a mechanism for controlling axial length growth.

Primary goals:

In a randomized 18 months prospective 1:1 study of a group of Danish children to:

1. Investigate if nightly wear of OKL (DreamliteR, Procornea, Nederlands) may reduce the progression of childhood myopia (change in axial length) when compared to a control group using SVS.
2. Investigate safety (Efron score) in the use of OKL.
3. Compare children's quality of life impact of refractive correction (questionnaire) using OKL and glasses.
4. Identify possible predictors for progression of myopia (AC/A ratio, peripheral defocus and higher order aberrations).

Hypothesis:

* Nightly wear of OKL reduces the progression of childhood myopia in Danish children.
* Use of OKL is safe, with no sight threatening complications during 18 months of nightly treatment.
* Children using OKL experience a higher quality of life impact of refractive correction compared to children wearing SVS.
* Response AC/A ratio is positively correlated to progression of childhood myopia.
* Use of OKL induce changes in corneal topography resulting in (1) decreased peripheral defocus (2) increased number of higher order aberrations. Progression in childhood myopia is associated to changes in peripheral defocus and higher order aberrations.

Design:

A 18-month randomized prospective 1:1 study of progression of myopia in a group of Danish children wearing OKL nightly (n=30) compared to a control group wearing SVS (n=30).

Children randomized to OKL will be examined at BL and day 3 and 7 as well as month 1, 3, 6, 9, 12, 15, and 18 after the start of treatment with OKL (T0).

Children randomized to SVS will be examined at BL and month 6, 12 and 18 after receiving new glasses with optimal prescription (T0).

Examination:

* Best corrected (using "push plus" refraction principle) ETDRS visual acuity: The OKL group (2-4 hours after lens removal) at BL and day 3 and 7 as well as month 1, 3, 6, 9, 12, 15, and 18 after T0. The SVS group at BL and month 6, 12 and 18 after T0.
* Grading contact lens complications (Efron Grading Scale for Contact Lens Complications) for the OKL group at day 3 and 7 as well as month 1, 3, 6, 9,12, 15, and 18 after T0.
* Dynamic auto-refraction (Shin-Nippon SRW-5000, Kagawa, Japan) for both groups at a distance of 40 cm in primary gaze as well as 5, 10, 20 and 30 degrees eccentric to the nasal and temporal retina in the horizontal meridian at BL and month 6, 12 and 18 after T0.
* Measurements of convergence for both groups at a distance of 40 cm and 6 meter using the Eye-Link 1000 (SR Research, Ontario, Canada) at BL and month 6, 12 and 18 after T0.
* Cycloplegic auto-refraction at BL, 6, 12, and 18 months (Topcon KR-800, Topcon Europe Medical, Capelle aan den Ijss, Nederlands).
* Axial length measurements (Lensstar, LS900, Carl Zeiss, Haag-Streit, Koeniz, Switzerland) at BL, 6, 12 and 18 months after T0 for both patients groups.
* Pentacam (Oculus, Wetzlar, Germany) for the OKL group at BL, T0, day 3, 7 as well as month 1, 3, 6, 9, 12, 15, and 18 after T0 (measurements obtained 2-4 hours after lens removal). For the group wearing SVS at BL, and month 6, 12 and 18 after T0.
* Pediatric Refractive Error Profile 2 (questionnaire) will be performed at 12 month for both patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Myopia -0.5 to -4.75 dioptries spherical in one or both eyes.
* Regular astigmatism ≤ -2.5 diopters in one or both eyes.
* Age 6 ≥ 12 years.
* Anisometropia < 1.5 D spherical equivalent.
* Best corrected visual acuity of 0.1 logMAR or better in both eyes.
* Acceptance of treatment randomization.

Exclusion Criteria:

* Manifest or latent squint.
* Contraindications to the use of OKL comprising keratoconus, allergic conjunctivitis and keratoconjunctivitis sicca.
* Previous eye surgery.
* Chronic eye disease demanding daily use of eye drops.
* Non-compliance to eye examinations (unstable fixation or intolerance to OKL).
* One or both parents being ethnical Asian, African, Hispanic or Spanish.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Progression of myopia defined as change in axial length 18 months after start of intervention | Follow up to 18 months

SECONDARY OUTCOMES:
Quality of life comparison between myopic children wearing glasses and orthokeratology lenses using the Pediatric Refractive Error Profile 2 Questionnaire | Follow up to 18 months
Safety evaluation by Efron scores for orthokeratology lenses | Follow up to 18 months
Accommodation and higher-order aberrations | Follow up to 18 months
  Median change in dynamic AC/A ratio and higher-order aberrations from BL to 18 months in myopic children wearing orthokeratology lenses and single-vision glasses

CONTACTS AND LOCATIONS:
Locations (1):
- Vejle Hospital, Vejle, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD is not to be shared with other researchers.

REFERENCES:
- [Derived] Cerullo C, Moller F, Ewan R, Norgaard B, Jakobsen TM. Vision-related quality of life in children: Cross-cultural adaptation and test-retest reliability of the Danish version of the paediatric refractive error profile 2. Acta Ophthalmol. 2024 Sep;102(6):e970-e983. doi: 10.1111/aos.16685. Epub 2024 Apr 13. PMID 38613420